CLINICAL TRIAL: NCT00390442
Title: Effect of Continuous Positive Airway Pressure as a First Line Therapy in Out-of-Hospital Management of Severe Cardiogenic Pulmonary Edema
Brief Title: Out-of-Hospital CPAP for Severe Cardiogenic Pulmonary Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hopital Lariboisière (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AOM03073, P030428, ENR20040504
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2006-10-19 (Estimated); Status verified 2006-10

CONDITIONS: Cardiogenic Pulmonary Edema
Keywords: cardiogenic pulmonary edema; non invasive ventilation; CPAP
MeSH Terms: interventions — Continuous Positive Airway Pressure

INTERVENTIONS:
Device: continuous positive airway pressure

SUMMARY:
In cardiogenic pulmonary edema, Continuous Positive Airway Pressure (CPAP) added to medical treatment improves outcome. The present study was designed to assess the benefit of CPAP as a first line treatment of cardiogenic pulmonary edema in the out-of-hospital environment.

DETAILED DESCRIPTION:
Cardiogenic pulmonary edema (CPE) is a frequent presenting process for acute out-of-hospital practice. Acute left heart failure may occur from a variety of processes that rapidly deteriorates to this generalized cardiopulmonary disorder. The classical treatment of out-of-hospital CPE includes supplemental oxygen, vasodilators, loop diuretics, and morphine. If not effective, or because of the associated respiratory depression, tracheal intubation and mechanical ventilation are often needed, which, by themselves are associated with a worse prognosis. Continuous positive airway pressure (CPAP) has been proposed as an alternative to mechanical ventilation in CPE. This technique not only improves alveolar recruitment and decreases the work of breathing 4 but also reduces left ventricular afterload, and both right and left ventricular preload. The overall effect of CPAP in the acute management of CPE is to improve cardio-respiratory function and sustained tissue oxygenation. Furthermore, the combination of CPAP with medical treatment in patients with CPE significantly reduces the need for intubation and improves the outcome.

Unfortunately, very limited data are available on the effects of CPAP in the out-of-hospital practice. Thus, we tested the potential benefit of immediate use of CPAP alone in comparison with pharmacological therapy in treatment of CPE in the acute out-of-hospital environment.

The protocol lasts 45 minutes, divided into 3 periods of 15 minutes. Patients with severe pulmonary edema are randomly assigned in 2 groups: 1/ "Early CPAP" (n=63): CPAP alone (T0-T15); CPAP + medical treatment (T15-T30); medical treatment alone (T30-T45); 2/ "Late CPAP" (n=61): medical treatment alone (T0-T15); medical treatment + CPAP (T15-T30); medical treatment alone (T30-T45). Primary endpoint : effect of early CPAP on a dyspnea clinical score and on arterial blood gases. Secondary endpoints : incidence of tracheal intubation, inotropic support, and in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical symptoms of acute pulmonary edema such as orthopnea, diffuse crackles without evidence of pulmonary aspiration or infection, percutaneous oxygen saturation  90% despite supplemental oxygen therapy (15 L.min-1) provided by the first responders were included in the study.

Exclusion Criteria:

* patients with a history of chronic obstructive pulmonary disease, asthma, severe stenotic valvular disease, or if they had cardiovascular collapse or an impaired level of consciousness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Primary endpoint : effect of early CPAP on a dyspnea clinical score and on arterial blood gases.

SECONDARY OUTCOMES:
Secondary endpoints :
incidence of tracheal intubation,
inotropic support,
in-hospital mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Plaisance, MD, PhD, Professor, Principal Investigator — Lariboisière Hospital
Locations (1):
- Lariboisiere University Hospital, Paris, France